CLINICAL TRIAL: NCT04442269
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Efficacy and Safety of Dupilumab in Patients With Allergic Bronchopulmonary Aspergillosis
Brief Title: Investigating Treatment With Dupilumab in Patients With Allergic Bronchopulmonary Aspergillosis (ABPA) (LIBERTY ABPA AIRED)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R668-ABPA-1923; 2019-002619-24 (EudraCT Number)
Record Dates: First submitted 2020-06-04; First posted 2020-06-22 (Actual); Results first posted 2024-08-21 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Allergic Bronchopulmonary Aspergillosis
MeSH Terms: conditions — Aspergillosis, Allergic Bronchopulmonary | interventions — dupilumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- dupilumab (Experimental): Loading subcutaneous (SC) dose on day 1, followed by SC dose, every two weeks (Q2W)
  Interventions: Drug: dupilumab
- Placebo (Experimental): Matching dupilumab without active substance
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: dupilumab — Single-use prefilled glass syringe administered by subcutaneous (SC) injection.
  Other Names: • DUPIXENT; • REGN668; • SAR231893
  Arms: dupilumab
Drug: Placebo — Matching placebo
  Arms: Placebo

SUMMARY:
The primary objective of the study is to evaluate the efficacy of dupilumab on lung function in participants with Allergic Bronchopulmonary Aspergillosis (ABPA).

The secondary objectives of the study are:

* To evaluate the effects of dupilumab on exacerbations in participants with ABPA
* To evaluate the effects of dupilumab on ABPA-related exacerbations
* To evaluate the effects of dupilumab on hospitalization/emergency department (ED)/urgent care visits in participants with ABPA
* To evaluate the effects of dupilumab on asthma control in participants with ABPA
* To evaluate the effects of dupilumab on health-related quality of life (HRQoL) in participants with ABPA
* To evaluate the effects of dupilumab on serum total immunoglobulin E (IgE) and Aspergillus-specific IgE concentrations
* To evaluate the effects of dupilumab on Fractional exhaled Nitric Oxide (FeNO) levels
* To evaluate safety and tolerability of dupilumab in participants with ABPA
* To evaluate dupilumab concentrations in serum and the incidence of anti-dupilumab antibodies in participants with ABPA

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of both ABPA and asthma
* On a maintenance therapy for their asthma with controller medication which must include inhaled corticosteroids (ICS) and may include 1 or more additional controller medications including a long-acting beta agonist (LABA), leukotriene receptor antagonist (LTRA), and/or long-acting muscarinic receptor antagonist (LAMA), etc for at least 12 weeks, with a stable dose and regimen with no change in the dose or frequency of administration for at least 4 weeks prior to the screening visit and between the screening and baseline/randomization visits
* For participants on OCS (oral corticosteroid): must be on a chronic stable dose (no change in the dose) of OCS of up to 10 mg/day (for participants taking daily corticosteroids) or up to 30 mg every alternate day (for participants taking alternate day corticosteroids) (prednisone/prednisolone or the equivalent) for at least 4 weeks prior to the screening visit and between the screening and the baseline/randomization visit
* Must have experienced ≥1 severe respiratory exacerbation requiring treatment with systemic corticosteroids or hospitalization or treatment in ED/urgent care within 12 months prior to the screening visit or must be receiving chronic stable low-dose OCS per above criteria

Key Exclusion Criteria:

* Weight less than 30.0 kilograms
* Current smoker or e-cigarette user, cessation of smoking or e-cigarette use within 6 months prior to randomization, or >=10 pack-years smoking history
* Post-bronchodilator FEV1 <30% predicted normal at screening
* Respiratory exacerbation requiring systemic corticosteroids within 4 weeks prior to screening and between screening and baseline visit (for patients on daily or alternate day OCS, exacerbation requiring at least double the maintenance dose of corticosteroids)
* Upper or lower respiratory tract infection within the 4 weeks prior to screening (visit 1) or between the screening and randomization visits
* Significant chronic pulmonary disease other than asthma complicated with ABPA (eg, physician-diagnosed bronchiectasis due to a condition other than ABPA; cystic fibrosis; sarcoidosis; interstitial lung disease not due to ABPA; chronic obstructive pulmonary disease [COPD] not due to ABPA; hypereosinophilic syndrome; etc), a diagnosed pulmonary or systemic disease associated with elevated peripheral eosinophil counts
* Diagnosis or suspected diagnosis of eosinophilic granulomatosis with polyangiitis (EGPA) (also called Churg-Strauss Syndrome)

NOTE: Other protocol defined inclusion / exclusion criteria applies.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2023-07-27 (Actual); Study Completion 2024-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (49):
- United States (13):
  - Regeneron Study Site, Birmingham, Alabama
  - Regeneron Study Site, Scottsdale, Arizona
  - Regeneron Study Site, Bakersfield, California
  - Regeneron Study Site, La Jolla, California
  - Regeneron Study Site, Los Angeles, California
  - Regeneron Study Site, Riverside, California
  - Regeneron Study Site, Boise, Idaho
  - Regeneron Study Site, Iowa City, Iowa
  - Regeneron Study Site, New York, New York
  - Regeneron Study Site, The Bronx, New York
  - Regeneron Study Site, Columbus, Ohio
  - Regeneron Study Site, DuBois, Pennsylvania
  - Regeneron Study Site, Philadelphia, Pennsylvania
- Bulgaria (4):
  - Regeneron Study Site, Haskovo
  - Regeneron Study Site, Razgrad
  - Regeneron Study Site, Smolyan
  - Regeneron Study Site, Sofia
- France (7):
  - Regeneron Study Site, Brest
  - Regeneron Study Site, Lyon
  - Regeneron Study Site, Marseille
  - Regeneron Study Site, Montpellier
  - Regeneron Study Site, Paris
  - Regeneron Study Site, Rennes
  - Regeneron Study Site, Tours
- Germany (3):
  - Regeneron Study Site, Leipzig, Saxony
  - Regeneron Study Site, Berlin
  - Regeneron Study Site, Frankfurt am Main
- Regeneron Study Site, Budapest, Hungary
- Japan (7):
  - Regeneron Study Site, Fukuyama
  - Regeneron Study Site, Kanagawa
  - Regeneron Study Site, Nagoya
  - Regeneron Study Site, Naka-gun
  - Regeneron Study Site, Sakai
  - Regeneron Study Site, Yanagawa
  - Regeneron Study Site, Yokohama
- Netherlands (5):
  - Regeneron Study Site, Amsterdam, North Holland
  - Regeneron Study Site, Arnhem
  - Regeneron Study Site, Breda
  - Regeneron Study Site, Eindhoven
  - Regeneron Study Site, Zutphen
- Poland (2):
  - Regeneron Study Site, Bialystok
  - Regeneron Study Site, Gdansk
- Romania (2):
  - Regeneron Study Site, Oradea, Bihor County
  - Regeneron Study Site, Brasov
- United Kingdom (5):
  - Regeneron Study Site, Leicester, England
  - Regeneron Study Site, Liverpool, England
  - Regeneron Study Site, London, England
  - Regeneron Study Site, Wythenshawe, England
  - Regeneron Study Site, Bradford, West Yorkshire

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Individual anonymized participant data will be considered for sharing once the indication has been approved by a regulatory body, if there is legal authority to share the data and there is not a reasonable likelihood of participant re-identification.
Access Criteria: Qualified researchers may request access to anonymized patient level data or aggregate study data when Regeneron has received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc) for the product and indication, has the legal authority to share the data, and has made the study results publicly available (eg, scientific publication, scientific conference, clinical trial registry).
URL: https://vivli.org/

REFERENCES:
- [Derived] Kao CC, Hanania NA, Parulekar AD. The impact of fungal allergic sensitization on asthma. Curr Opin Pulm Med. 2021 Jan;27(1):3-8. doi: 10.1097/MCP.0000000000000740. PMID 33027187
- See also: A Plain Language Summary is available on TrialSummaries.com — https://www.trialsummaries.com/

RESULTS

PARTICIPANT FLOW:
Groups:
- Dupilumab 300 mg Q2W: Subcutaneous (SC) dose every two weeks (Q2W)
Period: Overall Study
Arm/Group | Placebo | Dupilumab 300 mg Q2W
Started | 27 | 35
Completed | 20 | 29
Not Completed | 7 | 6
Not completed — Adverse Event | 1 | 0
Not completed — Death | 0 | 1
Not completed — Decision by the Investigator/Sponsor | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Protocol Deviation | 0 | 1
Not completed — Travel Limitations | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Dupilumab 300 mg Q2W | Total
Number analyzed (Participants) | 27 | 35 | 62
Age, Customized [Mean (Standard Deviation); unit: years] | 57.1 (14.38) | 61.2 (8.62) | 59.4 (11.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 22 | 39
  Male | 10 | 13 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 6
  Not Hispanic or Latino | 24 | 29 | 53
  Unknown or Not Reported | 1 | 2 | 3
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 25 | 28 | 53
  Asian | 1 | 4 | 5
  Other | 0 | 1 | 1
  Not Reported | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Pre-bronchodilator Forced Expiratory Volume in 1 Second (FEV1) Compared to Placebo
Time Frame: At Week 24
Population: Randomized participants with available data for analysis in the statistical model
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 26 | 34
Liters | 0.002 (0.0558) | 0.203 (0.0482)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg Q2W; Test type: Superiority; p = 0.0022, Mixed Models Analysis; Mean Difference = 0.201, 95% CI 2-sided [0.0768 to 0.3256]

2. Secondary Outcome: Annualized Rate of ABPA-related Exacerbations
Description: Defined as severe respiratory exacerbations that are associated with a doubling of serum total Immunoglobulin E (IgE) from the prior pre-exacerbation value.
  Adjusted Rate: Negative Binomial Regression Model Unadjusted Rate: (Number of events)/(number of participant years)
Time Frame: Over the 24 to 52 Week Treatment Period
Population: The full analysis set (FAS) includes all randomized participants. It is based on the treatment allocated as randomized
Measure: Number; unit: Events per person-year
Arm/Group | Placebo | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 27 | 35
Events per person-year
  Adjusted Rate | NA [NA to NA] — Negative Binomial Regression Model did not converge. | NA [NA to NA] — Negative Binomial Regression Model did not converge.
  Unadjusted Rate | 0 [0 to 0] | 0 [0 to 0]

3. Secondary Outcome: Annualized Rate of Severe Respiratory Exacerbations
Description: Defined as new onset of symptoms or clinical worsening of respiratory symptoms requiring systemic corticosteroid treatment for ≥3 consecutive days; for participants who are on maintenance systemic corticosteroids, at least double the dose of maintenance systemic corticosteroids for ≥3 consecutive days (with or without antibiotic therapy if indicated)
  Adjusted Rate: Negative Binomial Regression Model Unadjusted Rate: (Number of events)/(number of participant years)
Time Frame: Over the 24 to 52 Week Treatment Period
Population: The full analysis set (FAS) includes all randomized participants. It is based on the treatment allocated as randomized
Measure: Number; unit: Events per person year
Arm/Group | Placebo | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 27 | 35
Events per person year
  Adjusted Rate | 1.551 | 0.695
  Unadjusted Rate | 0.943 | 0.545

4. Secondary Outcome: Annualized Rate of Severe Respiratory Exacerbations Requiring Either Hospitalization or Observation for >24 Hours in an ED/Urgent Care Facility
Description: Annualized rate of severe respiratory exacerbations requiring either hospitalization or observation for >24 hours in an emergency department/urgent care facility (events per person-year)
  Adjusted Rate: Negative Binomial Regression Model Unadjusted Rate: (Number of events)/(number of participant years)
Time Frame: Over the 24 to 52 Week Treatment Period
Population: The full analysis set (FAS) includes all randomized participants. It is based on the treatment allocated as randomized
Measure: Number; unit: Events per person year
Arm/Group | Placebo | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 27 | 35
Events per person year
  Adjusted Rate | NA — Negative Binomial Regression Model did not converge. | NA — Negative Binomial Regression Model did not converge.
  Unadjusted Rate | 0.041 | 0.128

5. Secondary Outcome: Change From Baseline in Asthma Control Questionnaire (ACQ)-5 Score
Description: ACQ is completed by patient to measure both the adequacy of asthma control and change in asthma control, which occurs either spontaneously or as a result of treatment. The ACQ-5 score is the mean of the first 5 questions, between 0 (totally controlled) and 6 (severely uncontrolled). A higher score indicates lower asthma control. Participants with a score below 1.0 reflect adequately controlled asthma and participants with scores above 1.0 reflect inadequately controlled asthma. The optimal cut-point score of 1.50 should be used to be confident that a patient has inadequately controlled asthma.
Time Frame: Over the 24 to 52 Week Treatment Period
Population: Number of randomized patients with a baseline measurement and at least one post-baseline measurement at the post-baseline time point of interest
Measure: Mean (Standard Deviation); unit: ACQ-5 Score
Arm/Group | Placebo | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 27 | 35
ACQ-5 Score
  Week 24: number analyzed (Participants) | 23 | 32
  Week 24 | -1.10 (1.102) | -1.24 (1.081)
  Week 36: number analyzed (Participants) | 22 | 29
  Week 36 | -0.81 (0.878) | -1.15 (1.208)
  Week 44: number analyzed (Participants) | 20 | 26
  Week 44 | -0.87 (1.233) | -1.01 (1.359)
  Week 52: number analyzed (Participants) | 16 | 27
  Week 52 | -0.84 (1.183) | -1.29 (1.241)

6. Secondary Outcome: Change From Baseline in St. George's Respiratory Questionnaire (SGRQ) Total Score
Description: SGRQ will be completed by the patient to measure and quantify health status in adult participants with chronic airflow limitation. Total score ranges from 0 to 100. Scores by dimension are calculated for three domains: Symptoms, Activity, and Impacts (Psychosocial). Lower score indicates better Quality of Life (QoL).
Time Frame: Over the 24 to 52 Week Treatment Period
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: SGRQ Total Score
Arm/Group | Placebo | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 27 | 35
SGRQ Total Score
  Week 12: number analyzed (Participants) | 22 | 34
  Week 12 | -9.463 (16.3993) | -17.956 (14.6184)
  Week 24: number analyzed (Participants) | 22 | 31
  Week 24 | -7.626 (14.5412) | -23.079 (15.9104)
  Week 36: number analyzed (Participants) | 21 | 29
  Week 36 | -8.796 (16.4257) | -20.178 (15.5266)
  Week 52: number analyzed (Participants) | 19 | 28
  Week 52 | -8.938 (15.3127) | -25.309 (20.1035)

7. Secondary Outcome: Percentage of Participants Achieving a Reduction in the SGRQ Total Score of 4 Points or Greater From Baseline
Description: as for outcome 6
Time Frame: Up to 52 Weeks
Population: Participants must have both the baseline and at least one post-baseline measurement at the given post-baseline time point to be included in the calculation of the proportion at the given post-baseline time point.
Measure: Number (95% Confidence Interval); unit: Percent
Arm/Group | Placebo | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 27 | 35
Percent
  Week 12: number analyzed (Participants) | 22 | 34
  Week 12 | 50.0 [30.72 to 69.28] | 85.3 [69.87 to 93.55]
  Week 24: number analyzed (Participants) | 22 | 31
  Week 24 | 63.6 [42.95 to 80.27] | 87.1 [71.15 to 94.87]
  Week 36: number analyzed (Participants) | 21 | 29
  Week 36 | 57.1 [36.55 to 75.53] | 86.2 [69.44 to 94.50]
  Week 52: number analyzed (Participants) | 19 | 28
  Week 52 | 68.4 [46.01 to 84.64] | 89.3 [72.80 to 96.29]

8. Secondary Outcome: Percent Change From Baseline in Total IgE in Serum
Time Frame: Over the 24 to 52 Week Treatment Period
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Placebo | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 27 | 35
Percent
  Week 24: number analyzed (Participants) | 24 | 32
  Week 24 | -0.665 (40.2236) | -47.245 (19.4110)
  Week 36: number analyzed (Participants) | 22 | 29
  Week 36 | -5.945 (27.6767) | -57.752 (18.0812)
  Week 52: number analyzed (Participants) | 21 | 28
  Week 52 | -2.767 (42.8914) | -62.175 (17.0285)

9. Secondary Outcome: Percent Change From Baseline in A Fumigatus-specific IgE in Serum
Time Frame: Over the 24 to 52 Week Treatment Period
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Placebo | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 27 | 35
Percent
  Week 24: number analyzed (Participants) | 23 | 32
  Week 24 | 0.099 (39.7612) | -39.859 (25.3095)
  Week 36: number analyzed (Participants) | 21 | 30
  Week 36 | 6.766 (39.9041) | -45.654 (26.7915)
  Week 52: number analyzed (Participants) | 21 | 27
  Week 52 | 12.618 (94.6306) | -49.126 (30.6790)

10. Secondary Outcome: Absolute Change From Baseline in Fractional Exhaled Nitric Oxide (FeNO)
Time Frame: Over the 24 to 52 Week Treatment Period
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ppb
Arm/Group | Placebo | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 27 | 35
ppb
  Week 24: number analyzed (Participants) | 20 | 26
  Week 24 | -4.80 (23.521) | -22.04 (38.410)
  Week 36: number analyzed (Participants) | 18 | 29
  Week 36 | 3.11 (20.571) | -21.48 (40.538)
  Week 44: number analyzed (Participants) | 21 | 28
  Week 44 | 1.38 (21.896) | -19.18 (37.122)
  Week 52: number analyzed (Participants) | 19 | 26
  Week 52 | -4.79 (27.634) | -19.04 (35.471)

11. Secondary Outcome: Percent Change From Baseline in Fractional Exhaled Nitric Oxide (FeNO)
Time Frame: Over the 24 to 52 Week Treatment Period
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Placebo | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 27 | 35
Percent
  Week 24: number analyzed (Participants) | 20 | 26
  Week 24 | 1.67 (44.069) | -29.91 (32.527)
  Week 36: number analyzed (Participants) | 18 | 29
  Week 36 | 19.80 (44.053) | -24.56 (43.975)
  Week 44: number analyzed (Participants) | 21 | 28
  Week 44 | 15.43 (54.887) | -19.83 (48.308)
  Week 52: number analyzed (Participants) | 19 | 26
  Week 52 | 2.55 (56.506) | -20.35 (48.100)

12. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) From Baseline
Time Frame: Through the end of the 52 Week Treatment Period
Population: The safety analysis set (SAF) includes all randomized participants who received any study drug; it is based on the treatment received
Measure: Number; unit: Participants with TEAEs
Arm/Group | Placebo | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 27 | 35
Participants with TEAEs | 22 | 30

13. Secondary Outcome: Number of Participants With Treatment-emergent Anti-drug Antibody (ADA) Responses and Titer Over Time
Time Frame: Up to 64 Weeks
Population: The Pharmacokinetic Analysis Set (PKAS) includes all randomized participants who received any study drug and who had at least one non-missing drug concentration result following the first dose of study drug. The PKAS is based on the treatment received rather than as randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 25 | 34
Participants
  TE & TB Maximum Titer Category Low (<1,000) | 0 | 1
  TE & TB Maximum Titer Category Moderate (1,000 to 10,000) | 0 | 0
  TE & TB Maximum Titer Category High (>10,000) | 0 | 0

14. Secondary Outcome: Concentrations of Functional Dupilumab in Serum by Treatment Regimen
Time Frame: Up to 64 Weeks
Population: Includes all randomized participants who received dupilumab and who had at least one non-missing dupilumab result following the first dose. The PKAS is based on the treatment received rather than as randomized.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 34
mg/L
  Week 0: number analyzed (Participants) | 33
  Week 0 | 0 (0)
  Week 12: number analyzed (Participants) | 31
  Week 12 | 63.8 (35.4)
  Week 24: number analyzed (Participants) | 33
  Week 24 | 86.5 (53.6)
  Week 52: number analyzed (Participants) | 32
  Week 52 | 82.2 (55.4)
  Week 64: number analyzed (Participants) | 29
  Week 64 | 1.67 (4.38)

ADVERSE EVENTS:
Time Frame: From Day 1 to EOS (End Of Study) visit ~(up to 64 weeks)
Arm/Group | Placebo | Dupilumab 300 mg Q2W
All-Cause Mortality (participants affected / at risk) | 1/27 | 1/35
Serious Adverse Events (participants affected / at risk) | 5/27 | 3/35
Other Adverse Events (participants affected / at risk) | 19/27 | 29/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=27) | Dupilumab 300 mg Q2W (N=35)
Influenza (Infections and infestations) | 0 (0) | 2 (2)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 2 (2)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchopulmonary aspergillosis allergic (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Trisomy 16 (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=27) | Dupilumab 300 mg Q2W (N=35)
COVID-19 (Infections and infestations) | 3 (3) | 6 (6)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 4 (6)
Urinary tract infection (Infections and infestations) | 0 (0) | 4 (6)
Acute sinusitis (Infections and infestations) | 2 (2) | 2 (2)
Bronchopulmonary aspergillosis allergic (Infections and infestations) | 0 (0) | 2 (5)
Conjunctivitis (Infections and infestations) | 0 (0) | 2 (3)
Cystitis (Infections and infestations) | 0 (0) | 2 (3)
Lower respiratory tract infection (Infections and infestations) | 2 (3) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1) | 2 (3)
Respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
Rhinitis (Infections and infestations) | 0 (0) | 2 (2)
Sinusitis (Infections and infestations) | 1 (1) | 2 (2)
Tooth infection (Infections and infestations) | 0 (0) | 2 (3)
Viral upper respiratory tract infection (Infections and infestations) | 1 (2) | 2 (2)
Respiratory tract infection bacterial (Infections and infestations) | 3 (3) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 4 (35)
Injection site pain (General disorders) | 1 (1) | 3 (3)
Injection site swelling (General disorders) | 0 (0) | 3 (6)
Asthenia (General disorders) | 3 (9) | 2 (2)
Influenza like illness (General disorders) | 0 (0) | 2 (2)
Malaise (General disorders) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 2 (3)
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 4 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (6)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 9 (22) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 8 (15)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 2 (3) | 6 (15)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 1 (1)
Blepharitis (Eye disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2023-03-24): https://cdn.clinicaltrials.gov/large-docs/69/NCT04442269/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-05): https://cdn.clinicaltrials.gov/large-docs/69/NCT04442269/SAP_001.pdf